CLINICAL TRIAL: NCT02993731
Title: A Phase III Study of BBI-608 Plus Nab-Paclitaxel With Gemcitabine in Adult Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: A Study of Napabucasin Plus Nab-Paclitaxel With Gemcitabine in Adult Patients With Metastatic Pancreatic Adenocarcinoma
Acronym: CanStem111P
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CanStem111P
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: Neoplasms; Neoplasms by Site; Digestive System Neoplasms; Endocrine Gland Neoplasms; Pancreatic Neoplasms; Adenocarcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Digestive System Diseases; Pancreatic Diseases; Endocrine System Diseases; Albumin-Bound Paclitaxel; Gemcitabine
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Neoplasms; Neoplasms by Site; Digestive System Neoplasms; Endocrine Gland Neoplasms; Pancreatic Neoplasms; Adenocarcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Digestive System Diseases; Pancreatic Diseases; Endocrine System Diseases | interventions — napabucasin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Napabucasin plus Nab-paclitaxel with Gemcitabine (Experimental): Patients randomized to this arm will receive napabucasin administered orally, twice daily in combination with weekly nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks.
  Interventions: Drug: Napabucasin; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Arm 2: Nab-paclitaxel with Gemcitabine (Active Comparator): Patients randomized to this arm will receive weekly nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks.
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Napabucasin — Napabucasin will be administered orally, twice daily, with doses separated by approximately 12 hours.
  Other Names: BBI-608; BBI608; BB608
  Arms: Arm 1: Napabucasin plus Nab-paclitaxel with Gemcitabine
Drug: Nab-paclitaxel — Nab-paclitaxel 125 mg/m^2 immediately followed by gemcitabine 1000 mg/m^2 will be administered on Days 1, 8 and 15 of every 28-day cycle via intravenous infusion.
  Other Names: Abraxane
Drug: Gemcitabine — Nab-paclitaxel 125 mg/m^2 immediately followed by gemcitabine 1000 mg/m^2 will be administered on Days 1, 8 and 15 of every 28-day cycle via intravenous infusion.
  Other Names: Gemzar

SUMMARY:
This is a randomized, open-label, multi-center, phase 3 study of napabucasin plus weekly nab-paclitaxel with gemcitabine versus weekly nab-paclitaxel with gemcitabine for adult patients with Metastatic Pancreatic Ductal Adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Written, signed consent for trial participation must be obtained from the patient appropriately in accordance with applicable International Conference on Harmonization (ICH) guidelines and local and regulatory requirements prior to the performance of any study specific procedure.
2. Must have histologically or cytologically confirmed advanced pancreatic ductal adenocarcinoma (PDAC) that is metastatic. The definitive diagnosis of metastatic PDAC will be made by integrating the histopathological data within the context of the clinical and radiographic data. Patients with islet cell neoplasms are excluded.
3. Must not have previously received chemotherapy or any investigational agent for the treatment of PDAC. A fluoropyrimidine or gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed for as long as last dose was administered > 6 months prior to randomization and no lingering toxicities are present.
4. Nab-paclitaxel with gemcitabine therapy is appropriate for the patient and recommended by the Investigator.
5. Patient has one or more metastatic tumors evaluable by CT scan with contrast (or MRI, if patient is allergic to CT contrast media) per RECIST 1.1. Imaging investigations including CT/MRI of chest/abdomen/pelvis or other scans as necessary to document all sites of disease must be performed within 14 days prior to randomization. Qualifying scans performed as part of standard of care prior to patient signature of the study informed consent will be acceptable as baseline scanning as long as scanning is performed < 14 days prior to randomization.
6. Must have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1, assessed within 14 days prior to randomization. Two observers qualified to perform assessment of the performance status will be required to perform this assessment. If discrepant, the one with the most deteriorated performance status will be considered true.
7. Must have life-expectancy of > 12 weeks.
8. Must be ≥ 18 years of age. Due to increased risk of sepsis in patients >80 years old, candidate patients in this age group should be thoroughly evaluated prior to study randomization to ensure they are fit to receive chemotherapy. In addition to all of the inclusion/exclusion criteria listed, clinical judgment should be used regarding patients' susceptibility to infection (including but not limited to presence of ascites or diabetes mellitus increasing risk of infection). Furthermore, the expected stability of their performance status while receiving repeat weekly chemotherapy cycles should be given special attention. Patients in this age group should not be randomized on the study should there be any hesitation on any of these considerations.
9. For male or female patients of child producing potential: Must agree to use contraception or take measures to avoid pregnancy during the study and for 180 days after the final dose of nab-paclitaxel and gemcitabine or for 30 days for female patients and for 90 days for male patients, after the final napabucasin dose if nab-paclitaxel and gemcitabine were not administered.
10. Women of child bearing potential (WOCBP) must have a negative serum or urine pregnancy test within 5 days prior to randomization.
11. Patient has adequate biological parameters as demonstrated by the following blood counts at baseline (obtained < 14 days prior to randomization; laboratory testing performed as part of standard of care prior to patient signature of informed consent for the study will be acceptable as baseline laboratory work as long as testing is performed < 14 days prior to randomization):

    1. Absolute neutrophil count (ANC) > 1.5 x 10^9/L
    2. Platelet count > 100,000/mm^3 (100 x 10^9/L). Must not have required transfusion of platelets within 1 week of baseline platelet count assessment.
    3. Hemoglobin (HgB) > 9 g/dL. Must not have required transfusion of red blood cells within 1 week of baseline Hgb assessment.
12. Patient has the following blood chemistry levels at baseline (obtained < 14 days prior to randomization; laboratory testing performed as part of standard of care prior to patient signature of informed consent for the study will be acceptable as baseline laboratory work as long as testing is performed < 14 days prior to randomization):

    1. AST (SGOT) and ALT (SGPT) ≤ 2.5 × institutional upper limit of normal (ULN) [≤ 5 × ULN in presence of liver metastases]
    2. Total bilirubin ≤ 1.5 x institutional ULN. If total bilirubin is > ULN and < 1.5 x ULN, it must be non-rising for at least 7 days.
    3. Serum creatinine within normal limits or calculated clearance > 60 mL/min/1.73 m^2 for patients with serum creatinine levels above or below the institutional normal value. If using creatinine clearance, actual body weight should be used for calculating creatinine clearance (eg. Using the Cockcroft-Gault formula). For patients with a Body Mass Index (BMI) > 30 kg/m^2, lean body weight should be used instead.
13. Patient not on anticoagulation has acceptable coagulation studies (obtained < 14 days prior to randomization; laboratory testing performed as part of standard of care prior to patient signature of informed consent for the study will be acceptable as baseline laboratory work as long as testing is performed < 14 days prior to randomization) as demonstrated by prothrombin time (PT) and partial thromboplastin time (PTT) below or within normal limits (+15%).

    Patients on anticoagulation must have coagulation values within the therapeutic range appropriate for the anti-coagulation indication.
14. Patient has no clinically significant abnormalities on urinalysis results (obtained < 14 days prior to randomization; laboratory testing performed as part of standard of care prior to patient signature of informed consent for the study will be acceptable as baseline laboratory work as long as testing is performed < 14 days prior to randomization).
15. Patient must have adequate nutritional status with Body Mass Index (BMI) > 18 kg/m^2 and body weight of > 40 kg with serum albumin > 3 g/dL.
16. Baseline laboratory evaluations must be done within 14 days prior to randomization and some must be repeated < 72 hours prior to randomization.
17. Patients requiring biliary stent placement must have biliary stent placed > 7 days prior to screening.
18. Pain symptoms should be stable (of tolerable Grade 2 or less).
19. Only patients with available archival tumor tissue must consent to provision of, and Investigator(s) must confirm access to and agree to submit a representative formalin fixed paraffin block of tumor tissue in order that the specific correlative marker assays (Correlative Studies) of this protocol may be conducted. Submission of the tissue does not have to occur prior to randomization. Where local center regulations prohibit submission of blocks of tumor tissue, two 2 mm cores of tumor from the block and 5-20 unstained slides of whole sections of representative tumor tissue are preferred. Where it is not possible to obtain two 2 mm cores of tumor from the block, 5-20 unstained slides of representative tumor tissue are also acceptable. Where no previously resected or biopsied tumor tissue exists or is available, on the approval of the Sponsor/designated CRO, the patient may still be considered eligible for the study.
20. Patient must consent to provision of a sample of blood in order that the specific correlative marker assays (Correlative Studies) may be conducted.
21. Patients must be accessible for treatment and follow up. Patients registered on this trial must receive protocol treatment and be followed at the participating center. This implies there must be reasonable geographical limits placed on patients being considered for this trial. Investigators must ensure that the patients randomized on this trial will be available for complete documentation of the treatment, response assessment, adverse events, and follow-up.
22. Protocol treatment is to begin within 2 calendar days of patient randomization for patients randomized to Arm 1. Patients randomized to Arm 2 must begin protocol treatment within 7 calendar days of randomization.
23. The patient is not receiving therapy in a concurrent clinical study and the patient agrees not to participate in other interventional clinical studies during their participation in this trial while on study treatment. Patients participating in surveys or observational studies are eligible to participate in this study.

Exclusion Criteria:

1. Patients with no evidence of metastatic disease as well as patients with a local recurrence following surgical resection of primary lesion.
2. Patient has experienced a decline in ECOG performance status between Baseline visit and within 72 hours prior to randomization.
3. Patient has a > 20% decrease in serum albumin level between Baseline visit and within 72 hours prior to randomization.
4. Patient has a > 10% decrease in weight between Baseline visit and within 72 hours prior to randomization.
5. Any prior anti-cancer chemotherapy, biologic or investigational therapy for PDAC.

   1. Patients receiving immunotherapy for non-cancer related treatment within < 4 weeks of first planned dose of study treatment will be excluded.
   2. A fluoropyrimidine or gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed for as long as last dose was administered > 6 months prior to randomization.
6. Major surgery within 4 weeks prior to randomization.
7. Any known brain or leptomeningeal metastases are excluded, even if treated.
8. Patients with clinically significant ascites or pleural effusions.
9. Women who are pregnant or breastfeeding. Women should not breastfeed while taking study treatment and for 4 weeks after the last dose of napabucasin or while undergoing treatment with nab-paclitaxel and gemcitabine and for 180 days after the last dose of nab-paclitaxel and gemcitabine.
10. Gastrointestinal disorder(s) which, in the opinion of the Principal Investigator, would significantly impede the absorption of an oral agent (e.g. active Crohn's disease, ulcerative colitis, extensive gastric and small intestine resection).
11. Unable or unwilling to swallow napabucasin capsules daily.
12. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements.

    1. History of cardiac disease: congestive heart failure (CHF) > New York Heart Association (NYHA) Class II; active coronary artery disease, myocardial infarction or coronary stenting within 6 months prior to randomization; unevaluated new onset angina within 3 months or unstable angina (angina symptoms at rest) or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
    2. Current uncontrolled hypertension (systolic blood pressure [BP] > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management) as well as prior history of hypertensive crisis or hypertensive encephalopathy.
    3. Significant vascular disease (e.g., aortic aneurysm, aortic dissection, symptomatic peripheral vascular disease including claudication, Leo Buerger's disease). Treated peripheral vascular disease that is stable for at least 6 months is allowed.
    4. Evidence of bleeding diathesis or clinically significant coagulopathy.
    5. Major surgical procedure (including open biopsy, significant traumatic injury, etc.) within 28 days, or anticipation of the need for major surgical procedure during the course of the study as well as minor surgical procedure (excluding placement of a vascular access device or bone marrow biopsy) within 7 days prior to randomization.
    6. Patients with clinically significant abnormalities on urinalysis at < 14 days prior to randomization.
    7. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to randomization.
    8. Ongoing serious, non-healing wound, ulcer, or bone fracture.
    9. Known infection with Human Immunodeficiency Virus (HIV), and/or active infection with hepatitis B, or hepatitis C.
    10. History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies.
    11. History of hemolytic-uremic syndrome.
    12. History of connective tissue disorders (eg, lupus, scleroderma, arteritis nodosa).
    13. Serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders that could compromise the patient's safety or the study data integrity.
13. Known hypersensitivity to gemcitabine, taxanes or any of their excipients, or the patient exhibits any of the events outlined in the Contraindications or Special Warnings and Precautions sections of the product or comparator Summary of Product Characteristics or Prescribing Information. Possible hypersensitivity to napabucasin or one of the excipients which include the azo dyes sunset yellow and allura red.
14. Neurosensory neuropathy > grade 2 at baseline.
15. Uncontrolled chronic diarrhea > grade 2 at baseline.
16. Patients being treated with Warfarin.
17. Patients with active, uncontrolled bacterial, viral or fungal infection(s) requiring systemic therapy
18. Patients with a history of other malignancies except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated by surgery alone or surgery plus radiotherapy with no evidence of disease continuously for > 5 years.
19. Any active disease condition which would render the protocol treatment dangerous or impair the ability of the patient to receive protocol therapy.
20. Any condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol, including patients with history of poor compliance or history of drug/alcohol abuse, or excessive alcohol beverage consumption that would interfere with the ability to comply with the study protocol. Patients planning to take a vacation for 14 or more consecutive days during the course of the study are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1134 (Actual)
Dates: Start 2016-12; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (267):
- United States (99):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Clearview Cancer Institute (CCI), Huntsville, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - St. Joseph Hospital of Orange, Orange, California
  - Torrance Health Association DBA Torrance Memorial, Redondo Beach, California
  - UC Davis, Sacramento, California
  - UCLA Medical Center Santa Monica Hematology And Oncology, Santa Monica, California
  - Kaiser Permanente - Vallejo Medical Center, Vallejo, California
  - Norwalk Hospital The C Anthony and Jean Whittingham Cancer Center, Norwalk, Connecticut
  - The C Anthony and Jean Whittingham Cancer Center, Norwalk, Connecticut
  - Helen F. Graham Cancer Center, Newark, Delaware
  - Georgetown University Medical Center (GUMC), Washington D.C., District of Columbia
  - Florida Cancer Specialists & Research Institute, Fort Myers, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - UF Health Cancer Center - Orlando Health, Orlando, Florida
  - Florida Cancer Specialists North, St. Petersburg, Florida
  - Florida Cancer Specialists East Region, Wellington, Florida
  - University Cancer & Blood Center, Athens, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Saint Alphonsus Health System, Boise, Idaho
  - NorthShore University Health Systems, Evanston, Illinois
  - Ingalls Cancer Research Center, Harvey, Illinois
  - Carle Cancer Center CCOP, Urbana, Illinois
  - Northwestern Medicine Regional Medical Group, Warrenville, Illinois
  - Parkview Physician Group (PPG), Fort Wayne, Indiana
  - Indiana University - Melvin and Bren Simon Cancer, Indianapolis, Indiana
  - Cotton O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Louisiana Hematology Oncology Associates (LHOA), Baton Rouge, Louisiana
  - Maine Center for Cancer Medicine - Scarborough, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - St. Luke's Hospital of Duluth, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro MN Clinical Oncology Research Consortium, Saint Louis Park, Minnesota
  - Jackson Oncology Associates, Jackson, Mississippi
  - University of Missouri - Ellis Fischel Cancer Cent, Columbia, Missouri
  - Saint Luke's Hospital, Kansas City, Missouri
  - HCA Midwest Division (Kansas City), Kansas City, Missouri
  - Mercy Clinic - Cancer & Hematology, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - UNM Cancer Research and Treatment Center, Albuquerque, New Mexico
  - San Juan Oncology Associates, Farmington, New Mexico
  - Basset Medical Center, Cooperstown, New York
  - North Shore Hematology Oncology Associates PC, East Setauket, New York
  - Hematology Oncology Associates of Central New York, East Syracuse, New York
  - Clinical Research Alliance, Lake Success, New York
  - Weill Cornell Medicine/ NewYork-Presbyterian, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University, Stony Brook, New York
  - Montefiore Cancer Center, The Bronx, New York
  - UNC Chapel Hill / Lineberger Comprehensive Cancer, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - Wake Forest Baptist Hospital, Winston-Salem, North Carolina
  - Gabrail Cancer Center (GCC) - Canton Facility, Canton, Ohio
  - Toledo Clinic Cancer Centers, Toledo, Ohio
  - Cancer Center of Southwest Oklahoma, Lawton, Oklahoma
  - Mercy Clinic Oncology and Hematology - McAuley, Oklahoma City, Oklahoma
  - Kaiser Permanente - Westside Medical Office, Hillsboro, Oregon
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center (FCCC) - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - GHS Cancer Institute, Greenville, South Carolina
  - Avera Medical Group, Sioux Falls, South Dakota
  - Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - SCRI - Tennessee Oncology, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Bon Secours Cancer Institute Medical Oncology, Midlothian, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - The Everett Clinic, Everett, Washington
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
  - West Virginia University Mary Babb Randolph Cancer Center (MBRCC), Morgantown, West Virginia
  - HSHS St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Ltd. - West Green Bay, Green Bay, Wisconsin
  - Aurora St. Luke's Medical Center - Vince Lombardi, Milwaukee, Wisconsin
- Australia (14):
  - Border Medical Oncology, East Albury, New South Wales
  - Macquarie University Hospital, Sydney, New South Wales
  - ICON Cancer Care, South Brisbane, South Australia
  - Cabrini Hospital, Malvern, Victoria
  - Blacktown Cancer and Haematology Centre, Blacktown
  - Border Medical Oncology, East Albury
  - The Austin Hospital, Heidelberg
  - Cabrini Hospital, Malvern
  - Sir Charles Gairdner Hospital, Nedlands
  - Prince of Wales Private Hospital, Randwick
  - ICON Cancer Care, South Brisbane
  - Macquarie University Hospital, Sydney
  - The Tweed Hospital, Tweed Heads
  - Sydney Adventist Hospital, Wahroonga
- Austria (5):
  - LKH Universitätsklinikum Graz, Graz
  - Landeskrankenhaus Medical University Innsbruck, Innsbruck
  - Landeskrankenhaus Feldkirch, Rankweil
  - Universitatsklinik far Innere Medizin III, Salzburg
  - Medical University Vienna, Vienna
- Belgium (7):
  - ULB Erasme, Brussels
  - Antwerp University Hospital, Edegem
  - UZ Ghent, Ghent
  - UZ Brussel, Jette
  - UZ Leuven, Leuven
  - CHU de Liege, Liège
  - CHU Dinant Godinne, Yvoir
- Canada (6):
  - Dr. Everett Chalmers Regional Hospital, Fredericton, New Brunswick
  - The Atlantic Clinical Cancer Research Unit (ACCRU), Halifax, Nova Scotia
  - Centre Hospitalier de St. Mary, Pointe-Claire, Quebec
  - Ciusssmcq, Trois-Rivières, Quebec
  - Cross Cancer Institute, Edmonton
  - University of Toronto - St. Michael's Hospital, Toronto
- China (26):
  - Beijing Cancer Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - The first hospital of jilin university, Changchun
  - Fujian Medical University Union Hospital, Fuzhou
  - Cancer Center of Guangzhou Medical University, Guangzhou
  - Guangdong General Hospital, Guangzhou
  - The First Affiliated Hospital Zhejiang University, Hangzhou
  - The Second Affiliated Hospital Zhejiang University, Hangzhou
  - Sir Run Shaw Hospital School of Medicine Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - The 81 Hospital of the Chinese Peoples Liberation Army, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - Huashan Hospital, Shanghai
  - Ren Ji Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - East Hospital of Tongji University, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - The First Affiliated Hospital of Xian Jiao Tong University, Xi'an
  - General Hospital of Ningxia Medical University, Yinchuan
  - Henan Cancer Hospital, Zhengzhou
- Czechia (5):
  - Onkologicke oddeleni, Benešov
  - Fakultni nemocnice Brno Interni hematoonkologicka klinika, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - Onkologické oddělení, Zlín
- France (11):
  - Hôpital Sud - CHU Amiens Picardie, Amiens
  - Hôpital Trousseau, CHRU de Tours, Chambray-lès-Tours
  - Hopital Edourard Herriot, Lyon
  - CHU-Hôtel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hopital Europeen Georges Pompidou, Paris
  - Poitiers University Hospital, Poitiers
  - Centre Eugene Marquis, Rennes
  - Clinique Saint Anne, Strasbourg
  - Hopital Civil de strasbourg, Strasbourg
  - Institute de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
- Germany (9):
  - Gesundheitszentrum St. Marien GmbH, Amberg
  - University Hospital Bonn, Bonn
  - Klinikum Chemnitz, Chemnitz
  - Krankenhaus Nordwest, Frankfurt am Main
  - Medizinische Hochschule, Hanover
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Universitätsmedizin Mannheim, Mannheim
  - Klinikum Bogenhausen, München
  - Klinikum Oldenburg AöR - UK für Innere Medizin, Oldenburg
- Italy (12):
  - Fondazione Poliambulanza, Brescia
  - Istituto Ricerca e la Cura del Cancro (IRCC), Candiolo
  - AOU Mater Domini, Catanzaro
  - Ospedale degli Infermi, Faenza
  - Santa Maria de Prato Hospital, Feltre
  - IRCCS - Studio e la Cura dei Tumori, Meldola
  - IRCCS Ospedale San Raffaele, Milan
  - AO SM Misericordia, Perugia
  - IRCCS Azienda Ospedaliera S.Maria Nuova, Reggio Emilia
  - Ospedale degli Infermi, Rimini
  - Dermatological Hospital San Lazzaro, Torino
  - ASST Settelaghi, Varese
- Japan (13):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR, Koto-Ku, Tokyo
  - Kyorin University Hopsital, Mitaka, Tokyo
  - Kyoto University Hospital, Kyoto
  - Osaka International Cancer Institute, Osaka
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
- Netherlands (4):
  - Medisch Centrum Leeuwarden (MCL), Leeuwarden
  - Zuyderland Medical Center, Sittard
  - University Medical Center Utrecht, Utrecht
  - Isala Ziekenhuis, Zwolle
- Poland (7):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Onkologii-Instytut im.M.Sklodowskiej-Curie, Gliwice
  - Przychodnia Lekarska KOMED, Konin
  - Klinika Chirurgii Onkologicznej, Lublin
  - Centrum Onkologii Ziemi Lubelskiej, Lublin
  - Samodzielny Publiczny Szpital Kliniczny, Poznan
  - Wojewodzki Szpital Zespolony, Torun
- Portugal (6):
  - Fundação Champalimaud, Lisbon
  - Hospital da Luz, Lisbon
  - Centro Hospitalar Lisboa Norte, Lisbon
  - Centro Hospitalar do Porto, E.P.E, Porto
  - IPO Porto Francisco Gentil, E.P.E., Porto
  - Centro Hospitalar Entre Douro e Vouga, Santa Maria da Feira
- Russia (16):
  - Kursk Regional Clinical Oncology Dispensary, Kislino, Kursk Oblast
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk
  - Republican Clinical Oncology Dispensary, Cheboksary
  - Llc Evimed, Chelyabinsk
  - Railway Clinical Hospital on station Chelyabinsk, Chelyabinsk
  - Republic Clinical Oncology Dispensary, Kazan'
  - N.N. Blokhin Russian Cancer Research Center, Moscow
  - Privolzhsk District Medical Center, Nizhny Novgorod
  - Budgetary Healthcare Institution of Omsk Region, Omsk
  - Orenburg Regional Clinical Oncology Dispensary, Orenburg
  - Pyatigorsk Oncology Dispensary, Pyatigorsk
  - St.Petersburg Medical Universitet n.a. I.P. Pavlov, Saint Petersburg
  - FSBI "Russian Research Centre of Radiology and Surgical Technologies", Saint Petersburg
  - City Clinical Oncology Dispensary, Saint Petersburg
  - Multi-type clinic 'REAVIZ', Samara
  - National Research Mordovia State University, Saransk
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (8):
  - Seoul national University Bundang Hospital, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (11):
  - Hospital Vall d´Hebron, Barcelona
  - Hospital Clínico y Provincial de Barcelona, Barcelona
  - (ICO) Hospital Duran i Reynals, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Fundacion Alcorcon, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - LinKou Chang Gung Memorial Hospital, Taoyuan District
- Ukraine (2):
  - Zaytsev Institute General and Urgent Surgery of National Academy Medical Science of Ukraine, Kharkiv
  - National Institute of Cancer, Kyiv

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1134 participants were randomized between February 2017 and February 2019.
Pre-assignment Details: Patients who died, withdrew consent to survival follow up or were lost to follow up were considered to have completed the study.
Groups:
- Napabucasin Plus Nab-paclitaxel With Gemcitabine: All participants who were randomized to Arm 1 to receive napabucasin administered orally, twice daily in combination with weekly nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks.
- Nab-paclitaxel With Gemcitabine: All participants who were randomized to Arm 2 to receive nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks.
Period: Overall Study
Arm/Group | Napabucasin Plus Nab-paclitaxel With Gemcitabine | Nab-paclitaxel With Gemcitabine
Started | 565 | 569
Completed | 464 | 464
Not Completed | 101 | 105
Not completed — Study Termination | 101 | 105

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Napabucasin Plus Nab-paclitaxel With Gemcitabine | Nab-paclitaxel With Gemcitabine | Total
Number analyzed (Participants) | 565 | 569 | 1134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 325 | 295 | 620
  >=65 years | 240 | 274 | 514
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240 | 263 | 503
  Male | 325 | 306 | 631
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 194 | 188 | 382
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 18 | 28
  White | 350 | 354 | 704
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: To assess the effect of napabucasin plus weekly nab-paclitaxel with gemcitabine versus weekly nab-paclitaxel with gemcitabine on the Overall Survival of patients with metastatic pancreatic ductal adenocarcinoma.
Time Frame: From 4 weeks after the patient has been off study therapy, every 4 weeks thereafter for 6 months, then every 3 months thereafter until death, the study closes or 3 years since treatment discontinuation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Napabucasin Plus Nab-paclitaxel With Gemcitabine | Nab-paclitaxel With Gemcitabine
Number analyzed (Participants) | 565 | 569
Months | 11.43 [10.51 to 12.19] | 11.73 [10.74 to 12.71]

2. Secondary Outcome: Progression Free Survival
Description: To assess the effect of napabucasin plus weekly nab-paclitaxel with gemcitabine versus weekly nab-paclitaxel with gemcitabine on the Progression Free Survival (PFS) of patients with metastatic pancreatic ductal adenocarcinoma. PFS is defined as the time from randomization to the first objective documentation of disease progression or death due to any cause.
Time Frame: From date of randomization, every 8 weeks, until the date of first documented objective disease progression, up to 36 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Napabucasin Plus Nab-paclitaxel With Gemcitabine | Nab-paclitaxel With Gemcitabine
Number analyzed (Participants) | 565 | 569
Months | 6.70 [5.68 to 7.26] | 6.08 [5.59 to 7.10]

3. Secondary Outcome: Disease Control Rate
Description: To assess the effect of napabucasin plus weekly nab-paclitaxel with gemcitabine versus weekly nab-paclitaxel with gemcitabine on the Disease Control Rate (DCR) of patients with metastatic pancreatic ductal adenocarcinoma. DCR is defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Time Frame: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Napabucasin Plus Nab-paclitaxel With Gemcitabine (Response Analysis Set): All participants who were randomized to Arm 1 to receive napabucasin administered orally, twice daily in combination with weekly nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks and had measurable disease per RECIST 1.1 at randomization.
- Nab-paclitaxel With Gemcitabine (Response Analysis Set): All participants who were randomized to Arm 2 to receive nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks and had measurable disease per RECIST 1.1 at randomization.
Arm/Group | Napabucasin Plus Nab-paclitaxel With Gemcitabine (Response Analysis Set) | Nab-paclitaxel With Gemcitabine (Response Analysis Set)
Number analyzed (Participants) | 556 | 559
Percentage of participants | 74 [71 to 78] | 76 [72 to 80]

4. Secondary Outcome: Overall Response Rate
Description: To assess the effect of napabucasin plus weekly nab-paclitaxel with gemcitabine versus weekly nab-paclitaxel with gemcitabine on the Overall Response Rate (ORR) of patients with metastatic pancreatic ductal adenocarcinoma. ORR is evaluated using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1).
Time Frame: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Napabucasin Plus Nab-paclitaxel With Gemcitabine (Response Analysis Set) | Nab-paclitaxel With Gemcitabine (Response Analysis Set)
Number analyzed (Participants) | 556 | 559
Percentage | 43 [39 to 47] | 43 [39 to 47]

5. Secondary Outcome: Number of Patients With Adverse Events
Description: All patients who have received at least one dose of napabucasin will be included in the safety analysis according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 4.0. The incidence of adverse events will be summarized by type of adverse event and severity.
Time Frame: Every 1-2 weeks from date of screening until protocol treatment discontinuation. Following permanent protocol treatment discontinuation, every 8 weeks, starting with the 4 week post-protocol treatment discontinuation visit, up to 36 months.
Measure: Count of Participants; unit: Participants
Groups:
- Napabucasin Plus Nab-paclitaxel With Gemcitabine (Safety Population): All participants who received at least 1 dose of napabucasin administered orally, twice daily in combination with weekly nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks.
- Nab-paclitaxel With Gemcitabine (Safety Population): All participants who received at least 1 dose of nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks.
Arm/Group | Napabucasin Plus Nab-paclitaxel With Gemcitabine (Safety Population) | Nab-paclitaxel With Gemcitabine (Safety Population)
Number analyzed (Participants) | 561 | 547
Participants | 560 | 543

6. Secondary Outcome: Mean Change From Baseline for Global Quality of Life (QoL) at 8 Weeks.
Description: QoL will be measured using the European Organization for Research and Treatment of Cancer Quality of Life questionnaire (EORTC-QLQ-C30) in patients with metastatic pancreatic ductal adenocarcinoma with napabucasin plus weekly nab-paclitaxel with gemcitabine versus weekly nab-paclitaxel with gemcitabine. EORTQ QLC-C30 is a questionnaire used to assess the overall quality of life in cancer patients - 28 questions use a 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions use a 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged and transformed to 0-100 scale; higher overall score = better quality of life.
Time Frame: 8 weeks
Population: Each patient has 1 score selected from questionnaires collected from scheduled and unscheduled visits per scale per analysis window. If a patient had more than 1 questionnaire collected in an analysis window, the one collected closest to the target day is selected; if questionnaires had same days from the target day, the later one is selected; if questionnaires collected from the same date, the worst one is selected.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Napabucasin Plus Nab-paclitaxel With Gemcitabine: All participants who were randomized to Arm 1 to receive napabucasin administered orally, twice daily in combination with weekly nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks, and had at least one valid assessment at each analysis window.
- Nab-paclitaxel With Gemcitabine: All participants who were randomized to Arm 2 to receive nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks, and had at least one valid assessment at each analysis window.
Arm/Group | Napabucasin Plus Nab-paclitaxel With Gemcitabine | Nab-paclitaxel With Gemcitabine
Number analyzed (Participants) | 420 | 430
Score on a scale | -1.63 (22.535) | -0.57 (23.402)

7. Other Pre Specified Outcome: Overall Survival in Biomarker Positive Patients
Description: To assess the effect of napabucasin plus weekly nab-paclitaxel with gemcitabine versus weekly nab-paclitaxel with gemcitabine on the Overall Survival of patients with metastatic pancreatic ductal adenocarcinoma in biomarker positive patients. This biomarker-positive sub-population is defined as those patients with phospho-STAT3 positivity based on immunohistochemical (IHC) staining of Formalin Fixed Paraffin Embedded (FFPE) tumor tissue.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Months
Groups:
- Napabucasin Plus Nab-paclitaxel With Gemcitabine (pSTAT3 Positive): All participants who were randomized to Arm 1 to receive napabucasin administered orally, twice daily in combination with weekly nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks and were assessed to have positive pSTAT3 status based on their biomarker data.
- Nab-paclitaxel With Gemcitabine (pSTAT3 Positive): All participants who were randomized to Arm 2 to receive nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks and were assessed to have positive pSTAT3 status based on their biomarker data.
Arm/Group | Napabucasin Plus Nab-paclitaxel With Gemcitabine (pSTAT3 Positive) | Nab-paclitaxel With Gemcitabine (pSTAT3 Positive)
Number analyzed (Participants) | 206 | 176
Months | 11.40 [10.02 to 12.42] | 10.78 [9.40 to 12.55]

8. Other Pre Specified Outcome: Progression Free Survival in Biomarker Positive Patients
Description: To assess the effect of napabucasin plus weekly nab-paclitaxel with gemcitabine versus weekly nab-paclitaxel with gemcitabine on the Progression Free Survival (PFS) of patients with metastatic pancreatic ductal adenocarcinoma in biomarker positive patients. PFS is defined as the time from randomization to the first objective documentation of disease progression or death due to any cause. This biomarker-positive sub-population is defined as those patients with phospho-STAT3 positivity based on immunohistochemical (IHC) staining of Formalin Fixed Paraffin Embedded (FFPE) tumor tissue.
Time Frame: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Napabucasin Plus Nab-paclitaxel With Gemcitabine (pSTAT3 Positive) | Nab-paclitaxel With Gemcitabine (pSTAT3 Positive)
Number analyzed (Participants) | 206 | 176
Months | 5.68 [5.49 to 7.39] | 5.82 [5.55 to 7.29]

9. Other Pre Specified Outcome: Disease Control Rate in Biomarker Positive Patients
Description: To assess the effect of napabucasin plus weekly nab-paclitaxel with gemcitabine versus weekly nab-paclitaxel with gemcitabine on the Disease Control Rate (DCR) of patients with metastatic pancreatic ductal adenocarcinoma in biomarker positive patients. DCR is evaluated using RECIST 1.1. This biomarker-positive sub-population is defined as those patients with phospho-STAT3 positivity based on immunohistochemical (IHC) staining of Formalin Fixed Paraffin Embedded (FFPE) tumor tissue.
Time Frame: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage
Groups:
- Napabucasin Plus Nab-paclitaxel With Gemcitabine (pSTAT3 Positive; Response Analysis Set): All participants who were randomized to Arm 1 to receive napabucasin administered orally, twice daily in combination with weekly nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks, were assessed to have positive pSTAT3 status based on their biomarker data and had measurable disease per RECIST 1.1 at randomization.
- Nab-paclitaxel With Gemcitabine (pSTAT3 Positive; Response Analysis Set): All participants who were randomized to Arm 2 to receive nab-paclitaxel and gemcitabine administered intravenously, once weekly, on 3 of every 4 weeks, were assessed to have positive pSTAT3 status based on their biomarker data and had measurable disease per RECIST 1.1 at randomization.
Arm/Group | Napabucasin Plus Nab-paclitaxel With Gemcitabine (pSTAT3 Positive; Response Analysis Set) | Nab-paclitaxel With Gemcitabine (pSTAT3 Positive; Response Analysis Set)
Number analyzed (Participants) | 203 | 173
Percentage | 75 [69 to 81] | 79 [72 to 84]

10. Other Pre Specified Outcome: Overall Response Rate in Biomarker Positive Patients
Description: To assess the effect of napabucasin plus weekly nab-paclitaxel with gemcitabine versus weekly nab-paclitaxel with gemcitabine on the Overall Response Rate (ORR) of patients with metastatic pancreatic ductal adenocarcinoma in biomarker positive patients. ORR is evaluated using RECIST 1.1. This biomarker-positive sub-population is defined as those patients with phospho-STAT3 positivity based on immunohistochemical (IHC) staining of Formalin Fixed Paraffin Embedded (FFPE) tumor tissue.
Time Frame: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Napabucasin Plus Nab-paclitaxel With Gemcitabine (pSTAT3 Positive; Response Analysis Set) | Nab-paclitaxel With Gemcitabine (pSTAT3 Positive; Response Analysis Set)
Number analyzed (Participants) | 203 | 173
Percentage | 42 [35 to 49] | 47 [40 to 55]

ADVERSE EVENTS:
Time Frame: Every 1-2 weeks from date of screening until protocol treatment discontinuation. Following permanent protocol treatment discontinuation, every 8 weeks, starting with the 4 week post-protocol treatment discontinuation visit, up to 36 months.
Arm/Group | Napabucasin Plus Nab-paclitaxel With Gemcitabine (Safety Population) | Nab-paclitaxel With Gemcitabine (Safety Population)
All-Cause Mortality (participants affected / at risk) | 419/561 | 400/547
Serious Adverse Events (participants affected / at risk) | 330/561 | 273/547
Other Adverse Events (participants affected / at risk) | 560/561 | 543/547
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Napabucasin Plus Nab-paclitaxel With Gemcitabine (Safety Population) (N=561) | Nab-paclitaxel With Gemcitabine (Safety Population) (N=547)
Abdominal pain (Gastrointestinal disorders) | 30 | 21
Vomiting (Gastrointestinal disorders) | 27 | 12
Diarrhoea (Gastrointestinal disorders) | 23 | 17
Nausea (Gastrointestinal disorders) | 21 | 12
Constipation (Gastrointestinal disorders) | 6 | 4
Large intestinal obstruction (Gastrointestinal disorders) | 6 | 0
Colitis (Gastrointestinal disorders) | 5 | 4
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 2
Ascites (Gastrointestinal disorders) | 4 | 5
Intestinal obstruction (Gastrointestinal disorders) | 4 | 4
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 0
Duodenal obstruction (Gastrointestinal disorders) | 3 | 2
Ileus (Gastrointestinal disorders) | 3 | 7
Obstruction gastric (Gastrointestinal disorders) | 3 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 5
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 7
Haematemesis (Gastrointestinal disorders) | 2 | 1
Large intestine perforation (Gastrointestinal disorders) | 2 | 1
Mechanical ileus (Gastrointestinal disorders) | 2 | 0
Melaena (Gastrointestinal disorders) | 2 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Malignant bowel obstruction (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Splenic artery aneurysm (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Truncus coeliacus thrombosis (Gastrointestinal disorders) | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 23 | 18
Pneumonia (Infections and infestations) | 14 | 21
Biliary tract infection (Infections and infestations) | 11 | 1
Cellulitis (Infections and infestations) | 11 | 7
Urinary tract infection (Infections and infestations) | 10 | 7
Bacteraemia (Infections and infestations) | 6 | 3
Septic shock (Infections and infestations) | 5 | 5
Diverticulitis (Infections and infestations) | 4 | 1
Infection (Infections and infestations) | 4 | 2
Liver abscess (Infections and infestations) | 4 | 8
Lung infection (Infections and infestations) | 4 | 3
Clostridium difficile colitis (Infections and infestations) | 3 | 0
Clostridium difficile infection (Infections and infestations) | 3 | 0
Anal abscess (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 2 | 2
Enterocolitis infectious (Infections and infestations) | 2 | 0
Peritonitis (Infections and infestations) | 2 | 3
Pyelonephritis (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 1
Anal infection (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Central nervous system infection (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Escherichia pyelonephritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Hepatic infection (Infections and infestations) | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Perihepatic abscess (Infections and infestations) | 1 | 0
Pneumonia chlamydial (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2
Escherichia sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pancreatic abscess (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1
Prostate infection (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 2
Skin infection (Infections and infestations) | 0 | 1
Splenic abscess (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Viral sepsis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Disease progression (General disorders) | 45 | 22
Pyrexia (General disorders) | 34 | 29
Asthenia (General disorders) | 10 | 11
Fatigue (General disorders) | 8 | 5
General physical health deterioration (General disorders) | 7 | 7
Chest pain (General disorders) | 3 | 2
Death (General disorders) | 3 | 2
Pain (General disorders) | 3 | 2
Chest discomfort (General disorders) | 1 | 0
Condition aggravated (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Device related thrombosis (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 1
Obstruction (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 22 | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 16
Neutropenia (Blood and lymphatic system disorders) | 8 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 4
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 2 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 3
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 | 0
Acquired haemophilia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 18 | 6
Decreased appetite (Metabolism and nutrition disorders) | 8 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 1
Failure to thrive (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 8 | 3
Cholangitis (Hepatobiliary disorders) | 7 | 15
Bile duct obstruction (Hepatobiliary disorders) | 4 | 7
Cholangitis acute (Hepatobiliary disorders) | 3 | 3
Bile duct stenosis (Hepatobiliary disorders) | 2 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 2
Portal vein thrombosis (Hepatobiliary disorders) | 2 | 0
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 1
Gallbladder perforation (Hepatobiliary disorders) | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 1
Haemobilia (Hepatobiliary disorders) | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1
Hypotension (Vascular disorders) | 5 | 2
Embolism (Vascular disorders) | 4 | 1
Capillary leak syndrome (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 3
Aneurysm ruptured (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 4
Embolism venous (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral venous disease (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 2
Trousseau's syndrome (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 4
Cerebral infarction (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Axonal neuropathy (Nervous system disorders) | 0 | 1
Cerebral thrombosis (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Lumbosacral plexopathy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Polyneuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 6 | 5
Neutrophil count decreased (Investigations) | 3 | 2
Platelet count decreased (Investigations) | 2 | 4
Bile output increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 3
Haemoglobin decreased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 1
Weight decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 3
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Influenza A virus test positive (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 0
Cardiac failure (Cardiac disorders) | 3 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 2 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 8 | 2
Renal failure (Renal and urinary disorders) | 4 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic complication (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Confusional state (Psychiatric disorders) | 3 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 3
Major depression (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 6
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Device occlusion (Product Issues) | 3 | 1
Device dislocation (Product Issues) | 1 | 1
Device extrusion (Product Issues) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Pancreaticoduodenectomy (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Napabucasin Plus Nab-paclitaxel With Gemcitabine (Safety Population) (N=561) | Nab-paclitaxel With Gemcitabine (Safety Population) (N=547)
Diarrhoea (Gastrointestinal disorders) | 410 | 213
Nausea (Gastrointestinal disorders) | 329 | 252
Vomiting (Gastrointestinal disorders) | 250 | 162
Abdominal pain (Gastrointestinal disorders) | 215 | 124
Constipation (Gastrointestinal disorders) | 194 | 209
Abdominal pain upper (Gastrointestinal disorders) | 70 | 46
Dyspepsia (Gastrointestinal disorders) | 47 | 34
Abdominal distension (Gastrointestinal disorders) | 44 | 32
Stomatitis (Gastrointestinal disorders) | 39 | 52
Ascites (Gastrointestinal disorders) | 29 | 31
Pyrexia (General disorders) | 211 | 203
Fatigue (General disorders) | 205 | 189
Oedema peripheral (General disorders) | 179 | 180
Asthenia (General disorders) | 143 | 137
Malaise (General disorders) | 48 | 30
Disease progression (General disorders) | 45 | 23
Pain (General disorders) | 33 | 34
Chills (General disorders) | 28 | 16
Anaemia (Blood and lymphatic system disorders) | 306 | 318
Neutropenia (Blood and lymphatic system disorders) | 145 | 165
Thrombocytopenia (Blood and lymphatic system disorders) | 105 | 126
Leukopenia (Blood and lymphatic system disorders) | 56 | 56
Decreased appetite (Metabolism and nutrition disorders) | 233 | 177
Hypoalbuminaemia (Metabolism and nutrition disorders) | 76 | 74
Hypokalaemia (Metabolism and nutrition disorders) | 65 | 55
Dehydration (Metabolism and nutrition disorders) | 61 | 37
Hyponatraemia (Metabolism and nutrition disorders) | 56 | 26
Hyperglycaemia (Metabolism and nutrition disorders) | 28 | 30
Neutrophil count decreased (Investigations) | 138 | 155
White blood cell count decreased (Investigations) | 120 | 137
Platelet count decreased (Investigations) | 111 | 143
Alanine aminotransferase increased (Investigations) | 92 | 93
Weight decreased (Investigations) | 91 | 69
Aspartate aminotransferase increased (Investigations) | 85 | 88
Blood alkaline phosphatase increased (Investigations) | 62 | 57
Blood bilirubin increased (Investigations) | 48 | 36
Gamma-glutamyltransferase increased (Investigations) | 28 | 30
Neuropathy peripheral (Nervous system disorders) | 125 | 133
Peripheral sensory neuropathy (Nervous system disorders) | 92 | 97
Dysgeusia (Nervous system disorders) | 82 | 84
Dizziness (Nervous system disorders) | 52 | 51
Headache (Nervous system disorders) | 49 | 43
Paraesthesia (Nervous system disorders) | 24 | 29
Alopecia (Skin and subcutaneous tissue disorders) | 212 | 210
Rash (Skin and subcutaneous tissue disorders) | 89 | 85
Pruritus (Skin and subcutaneous tissue disorders) | 48 | 51
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 29 | 32
Urinary tract infection (Infections and infestations) | 64 | 41
Upper respiratory tract infection (Infections and infestations) | 41 | 35
Pneumonia (Infections and infestations) | 31 | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 69 | 69
Cough (Respiratory, thoracic and mediastinal disorders) | 68 | 74
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 52 | 55
Back pain (Musculoskeletal and connective tissue disorders) | 68 | 65
Pain in extremity (Musculoskeletal and connective tissue disorders) | 43 | 39
Myalgia (Musculoskeletal and connective tissue disorders) | 41 | 44
Muscular weakness (Musculoskeletal and connective tissue disorders) | 30 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 51
Insomnia (Psychiatric disorders) | 62 | 70
Anxiety (Psychiatric disorders) | 38 | 28
Chromaturia (Renal and urinary disorders) | 50 | 7
Hypertension (Renal and urinary disorders) | 40 | 52
Hypotension (Renal and urinary disorders) | 23 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The primary author agrees to, prior to submitting a manuscript, abstract, or any other written/oral presentation describing the Results for publication/presentation, forward a copy to the Sponsor at least 45 days prior to their submission. The Sponsor may request an additional 30-day embargo. The Sponsor may require the primary author to delete any Confidential Information (other than the Clinical Results) and to require that any publication/presentation acknowledge the Sponsor's support.

DOCUMENTS (2):
  • Study Protocol (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/31/NCT02993731/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT02993731/SAP_001.pdf